CLINICAL TRIAL: NCT05478759
Title: Innovative Multimodal and Attention Training to Improve Emotion Communication in Veterans With TBI and PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4411-P
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Brain Injury; Post Traumatic Stress Disorder
Keywords: cognition; intervention; brain injury; emotion recognition; post traumatic stress disorder
MeSH Terms: conditions — Brain Injuries; Stress Disorders, Post-Traumatic | interventions — Motion Pictures

STUDY DESIGN:
Intervention Model Description: 20 Veterans with mTBI and PTSD will be randomized to multimodal and attention training or inactive control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMART and attention training (Experimental): Training to recognize affect and prosodic expressions of emotions combined with attention training.
  Interventions: Behavioral: Multimodal affect recognition training; Behavioral: Attention Training
- Brain Health Workshop and National Geographic Movies (Placebo Comparator): an inactive arm that matches sessions of intervention. BHW is education about the brain and cognition. National Geographic movies are viewed with the clinician and the participant answers questions about the movies.
  Interventions: Behavioral: Brain Health Workshop; Behavioral: National Geographic Movies

INTERVENTIONS:
Behavioral: Multimodal affect recognition training — 8 session, trains participants to recognize expression of emotion from a variety of stimuli, including dynamic stimuli (e.g., video instead of still pictures) and it employs both facial and vocal examples of emotion expression.
  Other Names: MMART
  Arms: MMART and attention training
Behavioral: Attention Training — computerized attention drill training
  Other Names: Brain HQ
  Arms: MMART and attention training
Behavioral: Brain Health Workshop — an education presentation on brain function and cognitive principles of learning with homework and quizzes on information covered.
  Other Names: BHW
  Arms: Brain Health Workshop and National Geographic Movies
Behavioral: National Geographic Movies — participant will watch movies and answer questions after
  Other Names: movies
  Arms: Brain Health Workshop and National Geographic Movies

SUMMARY:
Poor emotion recognition has been associated with poor quality of interpersonal relationships, loss of employment, behavioral problems, reduced social reintegration, social isolation and even suicide. Deficits in emotion recognition are common in traumatic brain injury (TBI) and in post-traumatic stress disorder (PTSD) but these deficits have not been well studied in Veterans with both mild TBI (mTBI) and PTSD. Currently there are no interventions for emotion recognition in Veterans with mTBI and PTSD, and interventions for severe TBI have lacked training of both facial and vocal emotion recognition. In a preliminary study of an innovative combination of facial and vocal modalities, a multimodal affect recognition training (MMART) showed promise but lacked attention training that is an essential component in recognizing emotions in our daily lives. Given the need to improve relationships and productivity in Veterans with mTBI and PTSD, a study is needed to determine the effectiveness of a MMART combined with attention training.

DETAILED DESCRIPTION:
Background. Deficits in emotion recognition are common in traumatic brain injury (TBI) and in post-traumatic stress disorder (PTSD) but these deficits have not been well studied in Veterans with both mild TBI (mTBI) and PTSD. Poor emotion recognition has been associated with poor quality of interpersonal relationships, loss of employment, behavioral problems, reduced social reintegration, social isolation and even suicide. Currently there are no interventions for emotion recognition deficits in Veterans with mTBI and PTSD, and interventions conducted in civilians with severe TBI have lacked training of both facial and vocal emotion recognition. In a preliminary study of an innovative combination of facial and vocal modalities, a multimodal affect recognition training (MMART) showed promise with significant improvement on the Florida Affect Battery (FAB) but lacked attention training that is an essential component in recognizing rapidly changing emotions in our everyday lives. Attention training using Brain HQ targets the required attention factors underlying emotion recognition. Given the need to improve relationships and productivity in Veterans with mTBI and PTSD, a randomized controlled trial is needed to determine the effectiveness of an innovative MMART combined with attention training to improve emotion recognition and everyday function.

Objective & Hypotheses. The objective of this randomized controlled trial is to determine the treatment effect of a MultiModal Affect Recognition Training (MMART) combined with attention training in Veterans with TBI/PTSD.

Hypothesis 1. MMART combined with attention training will significantly improve performance on tests of emotion recognition.

Hypothesis 2: Treatment gains will translate to functional activities. Primary measures. Florida Affect Battery (FAB) and the Community Reintegration in Service members (CRIS).

Secondary measures. Emotion Recognition Task (ERT), attention index of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), the Continuous Performance Task and the TBI Quality of Life (TBI-QOL) Ability to Participate in Social Roles and Activities.

Methods. 20 Veterans with mTBI and PTSD will be randomized to either the combined training or an inactive control group. Both groups will attend 16, one-hour in-person sessions over 8 weeks. Outcomes will be assessed at pre-, post-, 3 month-post-treatment. A linear regression will be used to determine significant improvement of the treatment group over the control group, with t-tests to demonstrate within group improvement. Effect size calculations will be used to determine the power needed for a future Merit proposal.

ELIGIBILITY:
Inclusion Criteria:

* Veterans with a diagnosis of mTBI and PTSD based on VA/Department of Defense guidelines.
* Emotion recognition deficit
* Attention deficit
* Corrected vision within normal limits
* Hearing within normal limits
* Fluent in English

Exclusion Criteria:

* premorbid history of schizophrenia
* bipolar disorder
* chronic medical or neurological diseases

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Florida Affect Battery (FAB), assessing change | week 1, week 11, week 22
  a standardized assessment of emotional affect and prosody recognition. normative scores range from 0-100 for each of the 12 subscales. Higher scores indicate better emotion recognition.
Community Reintegration of Service Members, assessing change | week 1, week 11, week 22
  Satisfaction questionnaire of community participation. Scores range from .43 to 2.15. 43 items with five rating options of 1-5. Higher scores indicate better community participation.

SECONDARY OUTCOMES:
Emotion Recognition Task, assessing change | week 1, week 11, week 22
  computerized assessment of emotional affect recognition. Correct responses range from 0-48 (higher scores indicate better emotion recognition) and correct response time ranges from 0 to infinity (lower scores indicate quicker response time).
Continuous Performance Task, assessing change | week 1, week 11, week 22
  computerized measures of sustained attention. 100 trials with accuracy ranging from 0-100 (higher scores indicate better attention) and response time from 0-60 (lower scores indicate quicker response time).
Attention Index of the Repeatable Battery for the Assessment of Neuropsychological Status, assessing change | week 1, week 11, week 22
  digit span and symbol digit to assess attention. Scaled scores range from 1-19, with higher scores indicating better attention.
Traumatic Brain injury quality of life | week 1, week 11, week 22
  quality of life questionnaire about community participation. 59 items with scores ranging from 59-295, with higher scores indicating better community participation.

CONTACTS AND LOCATIONS:
Overall Officials: Julia K. Waid-Ebbs, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets will be maintained locally and a de-identified, anonymized dataset will be made available in response to specific requests that meet the criteria described within this document and to data repositories i.e. FITBIR.
Supporting Information: Analytic Code
Time Frame: at closure of study and as long as FITBIR retains the data
Access Criteria: dependent on FITBIR criteria
URL: https://fitbir.nih.gov/